CLINICAL TRIAL: NCT06095063
Title: Effect of Deep Transcranial Magnetic Stimulation (dTMS) on Cognition in Older Adults With Subjective Cognitive Decline (SCD)
Brief Title: dTMS for Subjective Cognitive Decline
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rotman Research Institute at Baycrest (Other)
Collaborators: Brainsway (Industry); Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Linda Mah, MD, Clinician Scientist, Rotman Research Institute at Baycrest
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 21-01
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease; Subjective Cognitive Decline
MeSH Terms: conditions — Alzheimer Disease | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 20 sessions of dTMS and Cognitive Training (Experimental): Participants will receive dTMS followed by computerized cognitive training.
  dTMS: The motor threshold (MT) will be measured by delivering single stimulations to the motor cortex with gradually increased intensity. After defining the MT, the coil will be positioned anterior to the hot spot using the ruler on the participant's cap, and a dTMS session will be performed with the dosing of the stimulus intensity titrated slowly to approximately 120% of the motor threshold. On Day 1 of the treatment, stimulation will be delivered at an intensity ranging from 80% to 100% of the participant's MT depending on their initial tolerance to the stimulation. Stimulation intensity will then be slowly titrated by sequentially increasing the intensity by 10% over the remaining days of the first week until a maximum intensity of 120% of MT is achieved depending on the tolerability of the patient.
  Immediately following dTMS, participants will complete 20-30 minutes of cognitive training.
  Interventions: Device: Active Brainsway H7-Coil Deep TMS System; Other: Cognitive Training
- 20 sessions of sham/control stimulation and Cognitive Training (Sham Comparator): Participants will receive sham intervention followed by computerized cognitive training.
  The sham intervention consists of treatment with similar technical parameters which induce scalp sensations but do not penetrate into the brain.
  Immediately following dTMS, participants will complete 20-30 minutes of cognitive training.
  Interventions: Device: Sham Brainsway H7-Coil Deep TMS System; Other: Cognitive Training

INTERVENTIONS:
Device: Active Brainsway H7-Coil Deep TMS System — Deep Transcranial Magnetic Stimulation (dTMS) is a new form of TMS which allows direct stimulation of deeper neuronal pathways than the standard TMS. The H-coil is a novel dTMS coil designed to allow deeper brain stimulation without a significant increase of electric fields induced in superficial cortical regions. dTMS will be administered daily for 4 consecutive weeks.
  Arms: 20 sessions of dTMS and Cognitive Training
Device: Sham Brainsway H7-Coil Deep TMS System — In addition to the active H-coil, a sham coil is included in the system. The active and sham coils are connected to a control switch, which alternates between real and sham operation modes. The sham treatment will be administered daily for 4 consecutive weeks.
  Arms: 20 sessions of sham/control stimulation and Cognitive Training
Other: Cognitive Training — Cognitive training will be conducted using the BrainHQ software program.

SUMMARY:
Deep transcranial magnetic stimulation (dTMS) is a brain stimulation technique that involves generating a brief magnetic field in a coil that is placed on the scalp. The magnetic field passes through the skull and induces a weak electrical current in the brain that briefly activates neural circuits at the stimulation site. The Brainsway dTMS H7-Coil is able to target an area of the brain that has been shown in studies to be linked to greater resilience to cognitive decline. In this study, the investigators will combine dTMS with cognitive training in older adults with subjective cognitive decline (SCD) and examine the effect of this treatment on memory, other cognitive abilities, and mood. In addition, the investigators will examine the combined effects of dTMS and cognitive training on brain activity as measured using electroencephalography (EEG).

Approximately 30 older adults from ages 55 to 70 with SCD and a positive family history of Alzheimer's disease will be enrolled in this study.

DETAILED DESCRIPTION:
This study will examine the effects of combining cognitive remediation with neurostimulation using deep transcranial magnetic stimulation (dTMS) and the H7-coil to target the anterior cingulate cortex (ACC) in older adults at risk for developing Alzheimer's disease (AD). Thirty older adults with subjective cognitive decline (SCD) and a family history of AD will participate in a single-site randomized double-blind sham-controlled cross-over trial of dTMS of the ACC in conjunction with active cognitive remediation for both sham and dTMS interventions. The primary goal of the study is to establish the feasibility of dTMS and cognitive training as a means to improve cognitive abilities in SCD. Secondary goals are to obtain preliminary evidence of improvement in executive function and memory abilities following dTMS and cognitive training. This trial is a first step towards developing effective neurostimulation protocols to reduce cognitive decline in older adults at risk for developing AD.

ELIGIBILITY:
Inclusion Criteria:

* have a family history of late onset sporadic Alzheimer's disease (AD) as defined by having a first degree relative, living or deceased, with a probable or confirmed diagnosis of AD
* have subjective memory decline and concern about memory changes
* score 26 or higher on the Montreal Cognitive Assessment (MoCA)
* are willing to provide informed consent
* are able to follow the treatment schedule
* are stable on medications for 2 months and are not expected to change medication during the entire study period (if they are taking medications)
* have a satisfactory safety screening questionnaire for TMS
* have an informant/study partner who is able to complete study questionnaires regarding the participant

Exclusion Criteria:

* have a metal plate in their head, except in the mouth (such as an ear implant, implanted brain stimulators, aneurysm clips)
* have known increased pressure or a history of increased pressure in their brain, which may increase their risk for having seizures
* have a cardiac pacemaker
* have an implanted medication pump
* have a central venous line
* have a significant heart condition
* have current depression or a history of any psychotic disorder, bipolar disorder, eating disorder, obsessive compulsive disorder, post-traumatic stress disorder, or dementia other than AD
* have a history of substance abuse in the last 6 months
* have a history of stroke or other brain lesions
* have a personal history of epilepsy
* have a family history of epilepsy
* are a pregnant or breast-feeding woman
* have a history of abnormal MRI of the brain
* have significant hearing loss requiring use of hearing aids
* have untreated hypo- or hyper-thyroidism
* have TMS contraindications
* have unstable medical condition(s)
* regularly use benzodiazepines or other hypnotics within 2 weeks of randomization

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of scheduled treatment sessions that are attended by study participants | 19 weeks
  There are in total 20 sessions of dTMS intervention and 20 sessions of sham stimulation.

SECONDARY OUTCOMES:
Change in baseline memory performance on a neuropsychological battery | 19 weeks
  Memory score from the neuropsychological battery at baseline will be compared to 4 weeks of intervention and at 1-month follow-up.
Change in executive function performance on a neuropsychological battery | 19 weeks
  Executive function scores from the neuropsychological battery at baseline will be compared to 4 weeks of intervention and at 1-month follow-up.
Change in baseline in scores on the Geriatric Depression Scale (GDS). | 19 weeks
  GDS is a 15-item self-report scale that measures an elderly individual's mood. A score greater than 5 suggests that the individual may be depressed. Administration time is approximately 5 minutes.
  The scores at baseline will be compared to 4 weeks of intervention and at 1-month follow-up.
Change in baseline in scores on the Geriatric Anxiety Inventory (GAI). | 19 weeks
  The GAI is a 20-item self-report measure of anxiety developed for older adults. Administration time is approximately 5 minutes.
  The scores at baseline will be compared to 4 weeks of intervention and at 1-month follow-up.
Change in baseline in scores on the Neuropsychiatric Inventory Questionnaire (NPI-Q) | 19 weeks
  The NPI assesses dementia-related behavioural symptoms including delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, aberrant motor activity, night-time behavioural disturbances and appetite and eating abnormalities. Administration time is approximately 15 minutes.
  The scores at baseline will be compared to 4 weeks of intervention and at 1-month follow-up.
Change in slow wave and resting state activity | 17 weeks
  Measured with electroencephalography (EEG) following 4 weeks of intervention and at 1-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Mah, Principal Investigator — Baycrest Rotman Research Institute
Locations (1):
- Rotman Research Institute at Baycrest, Toronto, Ontario, Canada